CLINICAL TRIAL: NCT02398513
Title: Uncontrolled, Open-label, Non-randomized, Phase I Study to Investigate the Pharmacokinetics, Safety, Tolerability, and Efficacy of Regorafenib in Chinese Patients (China Mainland) With Advanced, Refractory Solid Tumors)
Brief Title: Regorafenib Phase I Study in Mainland Chinese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15823
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Stivarga, BAY73-4506) (Experimental): Patients enrolled in the study will start treatment with Regorafenib160 mg (given by four 40 mg tablets of Regorafenib) on Day 1 of the first week followed by 6 days off treatment (Cycle 0, single dosing period). After Cycle 0, Regorafenib 160 mg QD will be administered for 21 days, followed by 7 days off treatment. Treatment with Regorafenib will continue until the patient either progresses or meets one of the criteria for withdrawal prespecified in the study protocol.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Regorafenib 160 mg per oral

SUMMARY:
The primary objective of this study is to define the pharmacokinetic of Regorafenib administered orally as a single agent in Chinese patients with advance solid tumors.

The second objective include the evaluation of safety, tolerability, and efficacy of Chinese patents treated with Regorafenib

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (IC) obtained before any study specific procedure. Patients must be able to understand and be willing to sign the written informed consent
* Patients with histologically or cytologically confirmed,refractory,locally advanced or metastatic solid tumors who are not candidates for standard therapy or in whom the specific clinical indications for which Regorafenib is approved elsewhere in the world is considered an appropriate treatment option.
* Male or female Chinese patients living in China mainland >= 18 years
* Patients must have measurable or non-measurable disease according to RECIST, version 1.1
* Eastern Cooperative Oncology Group performance status (ECOG-PS 0 - 1)
* Body mass index (BMI) between 18 and 33 kg/m2 inclusive
* Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to dosing:

  * Platelet count >= 100,000/cubic millimeters (mm3), hemoglobin (Hb) >= 9 g/dl, leukocyte count > 3,000/mm3, absolute neutrophil count (ANC) >=1,500/mm3. Transfusion to meet the inclusion criteria will not be allowed.
  * Total bilirubin <= 1.5 x the upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3.0 x ULN (<= 5 x ULN for patients with liver involvement of their cancer)
  * Alkaline phosphatase limit <= 2.5 x ULN (<= 5 x ULN for patients whose cancer involves their liver and/or bone)
  * Lipase <= 1.5 x ULN
  * Serum creatinine <= 1.5 times ULN and estimated creatinine clearance (CLcr) >= 30 mL/min according to the Cockroft-Gault formula
* International normalized ratio (INR) <= 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) <= 1.5 x ULN. Patients being treated with anticoagulant, e.g. warfarin or heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care.
* Life expectancy of at least 3 months.
* Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment.

Exclusion Criteria:

* Prior treatment with Regorafenib
* Patients unable to swallow and retain oral medications
* Any other malignant disease treated < 3 years prior to study entry, except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Staging: Ta, Tis and T1)
* Symptomatic metastatic brain or meningeal tumors if the patient is < 6 months from definitive therapy, has evidence of tumor growth on an imaging study within 4 weeks prior to study entry and is on dexamethasone and not clinically stable with respect to the tumor at the time of study entry.
* Major surgical procedure, or significant traumatic injury within 28 days before start of study medication
* History of organ allograft
* Non-healing wound, ulcer, or bone fracture
* Uncontrolled hypertension (systolic blood pressure >150 millimeter of mercury (mmHg) or diastolic blood pressure >90 mmHg despite optimal medical management)
* Persistent proteinuria > 3.5 g/24 hours measured by urine protein-creatinine ratio from a random urine sample (>=Grade 3, NCI-CTCAE v 4.03).
* History of cardiac disease: congestive heart failure (CHF) >=NYHA (New York Heart Association) Class II. Active coronary artery disease unstable angina (angina symptoms at rest) or new-onset angina (within last 3 months) or myocardial infarction (MI) within past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum drug concentration in plasma) | Cycle 0 day 1, 0、0.5、1、2、3、4、6、8、12、24、36、48、72、96 hours
AUC(0-24) (AUC from time 0 h to time 24 h post-administration) | Cycle 0 day1, 0、0.5、1、2、3、4、6、8、12、24 hours
AUC(0-tlast) (AUC from time zero to the last data point>LLOQ) | Cycle0 day 1, 0、0.5、1、2、3、4、6、8、12、24、36、48、72、96 hours
Cmax.ss (Cmax at steady-state during a dosage interval) | Cycle 1 day 21, 0,0.5,1,2,3,4,6,8,12,24,36,48,72,96 hours
AUCt.ss (AUC for the dosing interval at steady-state) | cycle 1 day 21 0,0.5,1,2,3,4,6,8,12,24 hours

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 30 days
Tumor Response base don RECIST 1.1 criteria | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Shanghai, China